CLINICAL TRIAL: NCT06138626
Title: Anesthetic Fresh Gas Flow Alert Test
Brief Title: Test of Excessive Anesthetic Fresh Gas Flow Alerting in the Electronic Medical Record to Reduce Excessive Fresh Gas Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Daniel Gessner, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 63548
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alert active (Experimental): Anesthesia provider will see alert when fresh gas flow is excessive
  Interventions: Behavioral: Alert
- Alert inactive (No Intervention): Anesthesia provider will not see alert when fresh gas flow is excessive

INTERVENTIONS:
Behavioral: Alert — An alert that appears when anesthetic fresh gas flow is excessive
  Arms: Alert active

SUMMARY:
The primary objective of this quality improvement intervention is to test the efficacy of excessive fresh gas flow alerting in the electronic medical record for anesthesia providers.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia provider using electronic medical record at study site

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Mean change in average fresh gas flow from baseline at 90 days | Baseline, day 90
  Mean change in average total fresh gas flow, in liters per minute as recorded in the electronic medical record, when administering sevoflurane, averaged over 1 week at baseline and over 1 week at 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided